CLINICAL TRIAL: NCT06973512
Title: HABITS Study (Helping Addiction by Individualized Therapeutic Stimulation): Pilot Trial of Deep Brain Stimulation Guided By Stereoelectroencephalography for Treatment-Refractory Substance Use Disorders
Acronym: HABITS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Victor Tang, Addiction Psychiatrist and Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO Project ID: 4520
Record Dates: First submitted 2025-03-20; First posted 2025-05-15 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Addiction; Substance Use Disorder (SUD)
Keywords: addiction; substance use disorder; deep brain stimulation; stereoelectroencephalography; biomarker; electrophysiology
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): There will be one arm where everyone will receive DBS
  Interventions: Device: deep brain stimulation and stereoelectroencephalography

INTERVENTIONS:
Device: deep brain stimulation and stereoelectroencephalography — Deep brain stimulation guided by stereoelectroencephalography
  Other Names: deep brain stimulation; stereoelectroencephalography

SUMMARY:
Substance use disorder (SUD) or addiction to drugs/alcohol is a devastating disease. Over 40,000 overdose deaths have happened in Canada since 2016, 1 in 5 Canadians will have a SUD, and 70% of those with SUD continue to relapse, showing that we urgently need new treatments. The Helping Addiction by Individualized Therapeutic Stimulation (HABITS) Study is exploring deep brain stimulation (DBS) for people who have failed to quit harmful substances.

Over 250,000 people have received DBS, which is well-established for Parkinson's disease and has evidence of success in major depression and obsessive-compulsive disorder. DBS uses electricity to directly stimulate areas of the brain. However, for DBS to work effectively, it needs to be personalized to each individual, which will be pursued through stereoelectroencephalography (SEEG). DBS and SEEG are minimally invasive and reversible, with a low risk of side effects.

SEEG started over 70 years ago to find seizure location in the brain of children and adults with epilepsy. It now has been used for major depression and chronic pain to guide DBS. It involves inserting electrodes temporarily across critical brain areas and monitoring patients for several days. SEEG can provide an understanding of where addiction and craving are in the brain to guide the placement of DBS electrodes and device settings that are optimal for a person.

In the HABITS Study, 10 participants will receive DBS guided by SEEG and undergo 11 study visits. Individuals will first undergo detoxification with CAMH. Then, they will receive DBS and SEEG at Toronto Western Hospital, where they will stay for 1 to 2 weeks. Finally, they will be followed for a year, where they will receive standard psychiatric care.

SUD causes heavy burdens on individuals, families, healthcare systems, and society. The HABITS Study promises to personalize DBS to treat those who are struggling with severe addiction.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is a promising treatment for substance use disorder (SUD) as it can precisely target and modulate aberrant disease-implicated neural networks. It has the unique ability to directly stimulate deep brain structures and deliver long-term electrical stimulation. DBS is minimally invasive, reversible, and non-ablative, with a minor risk of serious adverse events. DBS is well-established for movement disorders, with over 250,000 procedures performed, and has FDA breakthrough device status for major depression and OCD. A 2023 review of DBS for SUD demonstrated its tremendous promise, with an average clinical improvement of 60%. But with only approximately 50 patients with SUD receiving DBS worldwide, more studies are urgently required.

Although one of the strengths of DBS is its ability to be individualized to patients, doing so is difficult. Two critical barriers of DBS are 1) identifying optimal DBS electrode targets as many brain areas are implicated in addiction and 2) selecting the correct stimulation settings as many are possible and detecting immediate effects of settings is difficult (in contrast to movement disorders, such as immediate tremor cessation).

In the HABITS Study, we aim to address these shortcomings by using stereoelectroencephalography (SEEG), a comprehensive drug craving provocation paradigm, and a newly developed AI driven analysis pipeline. SEEG has been in use since the 1960s and is the gold standard for medication-resistant epilepsy, which involves the implantation of intracranial electrodes across the brain, providing continuous electrophysiological recordings for multiple days to identify seizure location. SEEG has been recently used to guide DBS for major depression and chronic pain.

By leveraging SEEG to elucidate an objective, predictive biomarker of addiction (e.g., craving), this can be used to better guide DBS target selection and stimulation setting to improve the effectiveness of DBS for patients with SUD.

ELIGIBILITY:
Inclusion Criteria:

* Adult, Age 25-65
* Severe DSM-5 substance use disorder (SUD) as assessed by Structured Clinical Interview for DSM-5 (SCID-5)
* Treatment refractory as evidenced by non-response to an adequate trial of ≥2 evidence-based treatment modalities for their substance use disorder in the most recent 3 years of illness, as determined by the study clinical team
* Able to comply with study visit schedule and timeline
* Stable housing and reliable transportation
* Treatment-seeking (>7 on a 0-10 readiness ruler and open to the end-of-treatment outcome of abstinence)
* Capable of understanding and providing informed consent

Exclusion Criteria:

* Contraindications to neurosurgical interventions such as major medical co-morbidities, including uncontrolled hypertension, coagulopathy, severe diabetes, major organ system failure, active infection or history of implant-related infections, immunocompromised state, or malignancy with <5 years life expectancy
* Contraindications for MRI, including implanted metallic devices (e.g., non-MRI-safe cardiac pacemaker or neurostimulator; some artificial joints metal pins; surgical clips; or other implanted metal parts), or claustrophobia or discomfort in confined spaces
* Cardiac pacemaker/defibrillator, or other implanted stimulator
* Presence of epilepsy, stroke, or degenerative disorder of the nervous system
* Serious problems with literacy, vision, or hearing

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | From enrolment to study conclusion at 12 months.
  Adverse events associated with SEEG and DBS will be recorded.
Feasibility Assessed by Recruitment Rates and Protocol Adherence | Across 3 years of the anticipated study length.
  Feasibility will be evaluated through the following metrics:
  1. Recruitment Rates: yearly and total number of participants recruited.
  2. Protocol Adherence: percentage of completed study visits.

SECONDARY OUTCOMES:
Proportion of Negative Urine Toxicology for Primary Substance (%) Assed by Urinalysis | From enrolment to study conclusion at 12 months.
  Supervised urine specimens are collected and screened with a point-of-care immunoassay, followed by GC-MS confirmation. Negative is defined as analyte concentration below the laboratory cut-off for the participant's primary substance of use (e.g., < 300 ng/mL benzoylecgonine for cocaine). This outcome is the percentage of participants whose sample is negative at the Month 12 endpoint.
Change From Baseline in Days of Primary Substance Use Assessed by Timeline Follow-Back Self-Report | From enrolment to study conclusion at 12 months.
  Timeline Follow-Back (TLFB) is a validated calendar interview conducted by trained staff. At enrollment, participants report their substance use for the past 90 days, and then, post-intervention, they report the number of days they used their primary substance between each study visit until study conclusion at 12 months. The proportion of days of substance use compared to not using during the 90 days before enrolment is compared to the proportion of days used versus not post-operatively, where the metric is in percentage (%).
Self-Reported Substance Craving Assessed Using a 0-10 Visual Analog Scale | From enrolment to study conclusion at 12 months.
  Craving is assessed with a 0-10 Visual Analog Substance Craving Scale administered by trained research staff. Participants mark their current urge to use on RedCAP, where 0 = "no craving at all" and 10 = "strongest craving imaginable." This outcome is the change in score from baseline (Week 0) to the Month 12 endpoint (Week 52 ± 2 weeks). Scores range 0-10; lower values indicate reduced craving (better outcome).
Depressive Symptom Severity Assessed by Patient Health Questionnaire (PHQ-9) | From enrolment to study conclusion at 12 months.
  The 9-item Patient Health Questionnaire (PHQ-9) is a self-administered scale that rates the frequency of depressive symptoms over the past two weeks on a 4-point scale (0 = "Not at all" to 3 = "Nearly every day"). Total scores range 0-27; higher scores indicate more severe depression (cut-offs: 5 = mild, 10 = moderate, 15 = moderately severe, 20 = severe). The outcome is change in total score from baseline (Week 0) to the Month 12 endpoint (Week 52 ± 2 weeks). Negative values reflect clinical improvement.
Anxiety Symptom Severity Asssed by General Anxiety Disorder (GAD-7) | From enrolment to study conclusion at 12 months.
  The 7-item Generalized Anxiety Disorder Scale (GAD-7) is a self-administered questionnaire that rates the frequency of anxiety symptoms over the past two weeks on a 4-point scale (0 = "Not at all" to 3 = "Nearly every day"). Total scores range 0-21; higher scores indicate more severe anxiety (cut-offs: 5 = mild, 10 = moderate, 15 = severe). This outcome is the change in total score from baseline (Week 0) to the Month 12 endpoint (Week 52 ± 2 weeks). Negative values reflect clinical improvement.
Electrophysiology Activity Correlating with Craving Assed by Brain Recordings Using Deep Brain Stimulation Electrodes and Stereoelectroencephalography | From enrolment to 12 months.
  Stereoelectroencephalography and deep brain stimulation electrodes will be used to record electrophysiological signals from the brain, also known as local field potentials (LFP), during low and high craving periods post-operatively, to the end of the study. The electrophysiology correlate of craving will be assessed by selecting the LFP spectral feature that best discriminates high- vs low-craving states, which will be assessed by the feature with the highest area under the ROC curve (AUC) of a logistic-regression model.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health / Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
I am not familiar with the process